CLINICAL TRIAL: NCT06619691
Title: Hands on Fun Occupational Therapy Fine Motor Program
Brief Title: HOFOT Fine Motor Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-77
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Fine Motor Skills
Keywords: Preschool; fine motor program; fine motor skills; early childhood development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FIne Motor Program participants (Experimental): All enrolled participants will completed a fine motor intervention program over 8 weeks
  Interventions: Other: Fine motor skills

INTERVENTIONS:
Other: Fine motor skills — Only intervention

SUMMARY:
The aim of this study is to determine if an 8 week fine motor intervention program will lead to improve fine motor skills as measured by a standardized assessment (PDMS-3) in pre- and post-test.

DETAILED DESCRIPTION:
The aim of this study is to determine if an 8 week fine motor intervention program will lead to improve fine motor skills as measured by a standardized assessment (Peabody Developmental Motor Scale, 3rd edition) in pre- and post-test. The hypothesis is that a daily fine motor program will improve overall fine motor skills within 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* preschooler aged 3-5 years old enrolled in local preschool

Exclusion Criteria:

* None other than denial of parent consent or lack of child assent

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Peabody Developmental Motor Scale, 3rd Edition | 8 weeks
  Peabody Developmental Motor Scales, 3rd edition - Norm referenced and standardized assessment of fine motor skills for children ages birth-5.11

CONTACTS AND LOCATIONS:
Locations (1):
- Mercy University, Dobbs Ferry, New York, United States

IPD SHARING:
Plan to Share IPD: No